CLINICAL TRIAL: NCT03792893
Title: Comparison of Pulse Wave and Blood Pressure Parameters Before, During and After Exercise Ergometry in Healthy Female Subjects - a Randomized, Controlled, Single-blind Study
Brief Title: Comparison of Pulse Wave and Blood Pressure Measurements Before, During and After Ergometry in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: Universität Tübingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ERG_03
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Healthy Female Subjects
Keywords: Cardiovascular parameters; Blood Pressure; Pulse Wave; Ergometry; Somnotouch; BOSO-TM-2430

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher Blood Pressure (Experimental): BOSO-TM-2430 blood pressure cuff is applied to the upper arm with the previously determined higher systolic blood pressure. Intervention: Ergometry H
  Interventions: Other: Ergometry H
- Lower Blood Pressure (Experimental): BOSO-TM-2430 blood pressure cuff is applied to the upper arm with the previously determined lower systolic blood pressure. Intervention: Ergometry L
  Interventions: Other: Ergometry L

INTERVENTIONS:
Other: Ergometry H — After a pre-rest period of 12 minutes, the subjects are physically strained on the ergometer for 48 minutes (6 minutes loading phase followed by a 2-minute rest phase; 30 watts increase every 8 minutes up to a maximum load of 180 watts), followed by a 12-minute rest periodmaximum load of 180 watts), followed by a 15-minute post-rest period.
  BOSO-TM-2430 blood pressure cuff is applied to the upper arm with the previously determined higher systolic blood pressure (reference parameter).
  SOMNOtouchTM RESP and GeTeMed Vitaguard 3100 are accordingly applied to the arm with the previously determined lower systolic blood pressure.
  Arms: Higher Blood Pressure
Other: Ergometry L — After a pre-rest period of 12 minutes, the subjects are physically strained on the ergometer for 48 minutes (6 minutes loading phase followed by a 2-minute rest phase; 30 watts increase every 8 minutes up to a maximum load of 180 watts), followed by a 12-minute rest periodmaximum load of 180 watts), followed by a 15-minute post-rest period.
  BOSO-TM-2430 blood pressure cuff is applied to the upper arm with the previously determined lower systolic blood pressure (reference parameter).
  SOMNOtouchTM RESP and GeTeMed Vitaguard 3100 are accordingly applied to the arm with the previously determined higher systolic blood pressure.
  Arms: Lower Blood Pressure

SUMMARY:
The objective of this randomized, controlled single blind study is to compare pulse wave and blood pressure measurements before, during and after exercise ergometry in healthy female subjects.

DETAILED DESCRIPTION:
In a randomized single-blind study design the investigators explore how well blood pressure parameters calculated using a Pulse Transit Time-based method (device: SOMNOtouchTM RESP) match blood pressure parameters measured by a classic upper arm blood pressure cuff (BOSO-TM-2430 ) under standardized load conditions (ergometry).

In 30 healthy female subjects (age 18 - 40 years), cardiovascular parameters before, during and after a standardized load on a bicycle ergometer (half-lying position) are recorded with three different devices (BOSO-TM-2430 versus SOMNOtouchTM RESP versus GeTeMed Vitaguard 3100) and compared.

Primary outcome is the difference of the systolic blood pressure values between the devices BOSO-TM-2430 versus SOMNOtouchTM RESP during the three phases.

The BOSO-TM-2430 blood pressure cuff is applied randomized to the arm with the previously determined higher or lower systolic blood pressure mean difference. The subjects are blinded to the results of the measurements during ergometry.

After a pre-rest period of 12 minutes, the subjects are physically strained on the ergometer for 48 minutes (6 minutes loading phase followed by a 2-minute rest phase; 30 watts increase every 8 minutes up to a maximum load of 180 watts), followed by a 12-minute rest period. Measurements are taken every two minutes with the BOSO-TM-2430; data acquisition with the SOMNOtouchTM RESP and GeTeMed Vitaguard 3100 devices takes place continuously over a total duration of 72 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy at the time of the examinations
* Inconspicuous anamnesis regarding cardiovascular diseases and bronchial asthma
* resting heart rate 50 to 100 beats per minute
* Normal blood pressure or appropriately treated and controlled hypertension (systolic blood pressure ≤ 140 mmHg and diastolic blood pressure ≤ 90 mmHg)

Exclusion Criteria:

* Acute or chronic (especially cardiovascular) diseases, including cardiac arrhythmia and vegetative regulatory disorders (recorded via anamnesis)
* Taking allopathic medication: digitalis, beta blockers, antiarrhythmics
* Bronchial asthma (recorded by anamnesis)
* Alcohol abuse
* Heart diseases NYHA class IV
* Blood pressure side difference ≥ 10mmHg
* Fever (> 37,5°C)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Difference of the systolic blood pressure | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Primary outcome is the difference of the systolic blood pressure values between the devices BOSO-TM-2430 versus SOMNOtouchTM RESP during the three phases

SECONDARY OUTCOMES:
Diastolic Blood Pressure (SOMNOtouchTM RESP) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Diastolic Blood Pressure (mm Hg) measured with the SOMNOtouchTM RESP device
Mean Arterial Blood Pressure (SOMNOtouchTM RESP) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Mean Arterial Blood Pressure (mm Hg) measured with the SOMNOtouchTM RESP device
Pulse Pressure (SOMNOtouchTM RESP) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Pulse Pressure (mm Hg) measured with the SOMNOtouchTM RESP device
Heartrate (SOMNOtouchTM RESP) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Heartrate (beats per minute, bpm) measured with the SOMNOtouchTM RESP device
Oxygen saturation (SpO2, SOMNOtouchTM RESP) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Oxygen saturation (% SpO2) measured with the SOMNOtouchTM RESP device
Pulse-Transit-Time (PTT, SOMNOtouchTM RESP) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Pulse-Transit-Time (PTT, ms) measured with the SOMNOtouchTM RESP device
Systolic Blood Pressure measured with the device BOSO-TM-2430 | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Systolic Blood Pressure (mmHg) measured with the BOSO-TM-2430 device
Diastolic Blood Pressure measured with the device BOSO-TM-2430 | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Diastolic Blood Pressure (mmHg) measured with the BOSO-TM-2430 device
Mean Arterial Blood Pressure measured with the device BOSO-TM-2430 | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Mean Arterial Blood Pressure (mmHg) measured with the BOSO-TM-2430 device
Pulse Pressure measured with the device BOSO-TM-2430 | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Pulse Pressure (mmHg) measured with the BOSO-TM-2430 device
Heartrate measured with the device BOSO-TM-2430 | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Heartrate (beats per minute, bpm) measured with the BOSO-TM-2430 device
Pulse Transit Time (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Pulse Transit Time (PTT, ms) measured with the GeTeMed Vitaguard 3100 device
Perfusion Index (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Perfusion Index (PI) measured with the GeTeMed Vitaguard 3100 device
Peak to Peak Time (PPT) (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Peak to Peak Time (PPT, ms) measured with the GeTeMed Vitaguard 3100 device
SlopeInW1 (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  SlopeInW1 measured with the GeTeMed Vitaguard 3100 device
SlopeInW2 (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  SlopeInW2 measured with the GeTeMed Vitaguard 3100 device
SlopeInW3 (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  SlopeInW3 measured with the GeTeMed Vitaguard 3100 device
SlopeInW4 (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  SlopeInW4 measured with the GeTeMed Vitaguard 3100 device
StiffnessIndex (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  StiffnessIndex measured with the GeTeMed Vitaguard 3100 device
ReflectionIndex (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  ReflectionIndex measured with the GeTeMed Vitaguard 3100 device
TimeTX (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  TimeTX (ms) measured with the GeTeMed Vitaguard 3100 device
TimeTY (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  TimeTY (ms) measured with the GeTeMed Vitaguard 3100 device
QuotTYTX (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  QuotTYTX measured with the GeTeMed Vitaguard 3100 device
AreaAX (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  AreaAX measured with the GeTeMed Vitaguard 3100 device
AreaAY (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  AreaAY measured with the GeTeMed Vitaguard 3100 device
QuotAYAX (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  QuotAYAX measured with the GeTeMed Vitaguard 3100 device
AreaAV (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  AreaAV measured with the GeTeMed Vitaguard 3100 device
AreaAW (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  AreaAW measured with the GeTeMed Vitaguard 3100 device
QuotAWAV (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  QuotAWAV measured with the GeTeMed Vitaguard 3100 device
QuotTVTW (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  QuotTVTW measured with the GeTeMed Vitaguard 3100 device
TimeTV (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  TimeTV (ms) measured with the GeTeMed Vitaguard 3100 device
TimeTW (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  TimeTW (ms) measured with the GeTeMed Vitaguard 3100 device
MinT1 (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Minimum of the pulse wave measured with the GeTeMed Vitaguard 3100 device at the beginning of the first peak
MinT2 (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Minimum of the pulse wave measured with the GeTeMed Vitaguard 3100 device at the beginning of the second peak
MaxT1 (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Maximum of the pulse wave measured with the GeTeMed Vitaguard 3100 device at the maximum of the first peak
MaxT2 (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Maximum of the pulse wave measured with the GeTeMed Vitaguard 3100 device at the maximum of the second peak
QuotHRRespRate (GeTeMed Vitaguard 3100) | Physiological parameters are measured continuously (SOMNOtouchTM RESP) and every 2 minutes (BOSO-TM-2430) for a total duration of 72 minutes
  Quotient of heart and respiratory rates measured with the GeTeMed Vitaguard 3100 device

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, MD, Study Director — ARCIM Institute, Im Haberschlai 7, 70794 Filderstadt, Germany
Locations (1):
- ARCIM Institute, Filderstadt, Baden-Wurttemberg, Germany